CLINICAL TRIAL: NCT03808753
Title: Mini Fluid chAlleNge and End-expiratory Occlusion Test and to Assess flUid responsiVEness in opeRating Room: an Open-label, Randomized Clinical Trial
Brief Title: Mini Fluid chAlleNge and End-expiratory Occlusion Test and to Assess flUid responsiVEness in opeRating Room
Acronym: MANEUVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Principal Investigator, Antonio Messina, ICU senior consultant, Humanitas Clinical and Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MANEUVER_1
Record Dates: First submitted 2019-01-15; First posted 2019-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Hemodynamic Instability; Anesthesia; Surgery
Keywords: Mini Fluid Challenge; End-expiratory occlusion test; Fluid responsiveness; Functional Hemodynamic Test

STUDY DESIGN:
Intervention Model Description: The study protocol was started during a period of intraoperative hemodynamic stability, as previously defined (i.e. change in mean arterial pressure of less than 10% during 5 minutes). The study protocol is was the following: 1) a set of measurements was recorded (T0) at a baseline ventilation of 7 ml/Kg and then the EEOT is performed by using the software function, "expiratory hold", to interrupt mechanical ventilation; 2) after one minute a set of measurements was recorded (T1); 3) the mFC is then performed; 4) a FC of overall 4 mL/Kg of crystalloid solution is infused over 9 minutes (T2). The attending anesthetist is allowed to interrupt the protocol at any stage for either hemodynamic instability or any other adverse effects requiring urgent treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment - hemodynamic tests: EEOT and mFC (Experimental): Interventions: all the enrolled patients will be tested using the EEOT and the mFC.
  Interventions: Diagnostic Test: End-expiratory occlusion test (EEOT); Other: mini fluid challenge (mFC)

INTERVENTIONS:
Diagnostic Test: End-expiratory occlusion test (EEOT) — The EEOT is performed by interrupting the mechanical ventilation for 30 seconds, by using and end-expiratory hold on the ventilator.
Other: mini fluid challenge (mFC) — The mFC is performed by injecting a first aliquot of 100 ml of crystalloid over 1 minute before completing the 4 ml/kg-FC over the residual 9 minutes.

SUMMARY:
End-expiratory occlusion test (EEOT) has been previously successfully tested in surgical patients, consisting of the interruption of the mechanical ventilation for 30 seconds, and in the evaluation of the changes in the SV.

The mini fluid challenge test (mFC) aims at testing the increase in SV after the rapid administration of a small aliquot of the predefined FC.

Both these test have been previously evaluated in small-sized studies and never compared each other.

DETAILED DESCRIPTION:
Targeted fluid therapy has received increasing attention in the management of patients showing acute circulatory failure in both intensive care unit (ICU) and operating room (OR), aiming at preventing both inadequate tissue blood flow and fluid overload [1]. In fact, unnecessary fluid administration can increase morbidity and mortality and length of hospital stay of critically ill and surgical patients [2-10].

Since the only physiological reason to give a fluid challenge (FC) is to increase the stroke volume (SV) [11-13] and this effect is obtained only in about 50% of ICU and OR patients [14, 15], a vast literature investigated the possibility of predict this effect before FC administration, but the issue remains extremely challenging [1, 13, 16-18]. Bedside clinical signs and pressure and static volumetric static variables, do not predict fluid responsiveness [17]. Moreover, several physiological factors affect the reliability of the ventilator-induced dynamic changes in pulse pressure and stroke volume [pulse pressure variation (PPV) and stroke volume (SV) variation (SVV), respectively], and their echographic surrogates, in a significant number of ICU and OR patients [19-22].

To overcome these limitations, the functional hemodynamic assessment (i.e. the assessment of the dynamic interactions of hemodynamic variables in response to a defined perturbation), of fluid responsiveness has gained in popularity [17, 18, 23]. A functional hemodynamic test (FHT) consist in a manoeuvre determining a sudden change in cardiac function and/or heart lung interaction, affecting the hemodynamics of fluid responders and non-responders to a different extent [17, 18, 23].

The FHT called passive leg raising (PLR) has been successfully used for assessing the fluid responsiveness in ICU patients since 2009 [24] and its reliability has been confirmed by three large meta-analyses [25-27]. However, the PLR is not usually practicable in the OR.

A lot of different FHTs have been proposed, as alternative to the PLR, in ICU and, more recently, OR. These tests could be basically subdivided in two groups. A subgroup of FHTs is based on sudden and brief variations of the mechanical ventilation to induce a change in right ventricle preload and/or after load and, as consequence, of left ventricle SV [24, 28]. Among these tests, the end-expiratory occlusion test (EEOT) has been previously successfully tested in surgical patients, consisting of the interruption of the mechanical ventilation for 30 seconds, and in the evaluation of the changes in the SV. A second subgroup aims at testing the increase in SV after the rapid administration of a small aliquot of the predefined FC [29, 30]. This test is called mini fluid challenge (mFC). Both these test have been previously evaluated in small-sized studies and never compared each other.

The primary aim of the present study is to compare the reliability of EEOT and mFC in predicting fluid responsiveness in patients undergoing general surgery.

ELIGIBILITY:
All elective adults (age > 18 years) consecutive patients scheduled for elective abdominal surgery requiring invasive arterial monitoring and scheduled in those operating rooms equipped with ventilators having an expiratory-hold function.

The preoperative exclusion criteria were 1) any recurrent cardiac arrhythmia; 2) known reduced left (ejection fraction < 30%) or right (systolic peak velocity of tricuspid annular motion < 0.17 m/s) ventricular systolic function; Body Mass Index > 35; 4) chronic obstructive pulmonary disease classified as GOLD ≥ 2. Once enrolled, the patient can be additionally excluded because of the occurrence of one of the following intraoperative conditions: 1) significant bleeding (more than 500 ml in ½ hour); 2) persistent and/or recurrent extrasystoles; 3) persistent low quality of the arterial signal despite optimization of the signal (see further).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
ROC curve calculation | 10 minutes
  Calculation of the area under the ROC curve considering the response to the fluid challenge test (considered as gold standard).

SECONDARY OUTCOMES:
ROC:Comparison of the areas under the ROC curve of each test (EEOT and mFC) | 10 minutes
  Comparison of the areas under the ROC curve of each test (EEOT and mFC)

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Humanitas Research Hospital, Rozzano, Milano
  - Careggi University Hospital, Florence, Tuscany
  - Maggiore della Carità University Hospital, Novara

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Messina A, Pelaia C, Bruni A, Garofalo E, Bonicolini E, Longhini F, Dellara E, Saderi L, Romagnoli S, Sotgiu G, Cecconi M, Navalesi P. Fluid Challenge During Anesthesia: A Systematic Review and Meta-analysis. Anesth Analg. 2018 Dec;127(6):1353-1364. doi: 10.1213/ANE.0000000000003834. PMID 30300177
- [Background] Pinsky MR. Functional hemodynamic monitoring. Crit Care Clin. 2015 Jan;31(1):89-111. doi: 10.1016/j.ccc.2014.08.005. PMID 25435480
- [Background] Muller L, Toumi M, Bousquet PJ, Riu-Poulenc B, Louart G, Candela D, Zoric L, Suehs C, de La Coussaye JE, Molinari N, Lefrant JY; AzuRea Group. An increase in aortic blood flow after an infusion of 100 ml colloid over 1 minute can predict fluid responsiveness: the mini-fluid challenge study. Anesthesiology. 2011 Sep;115(3):541-7. doi: 10.1097/ALN.0b013e318229a500. PMID 21792056
- [Background] Cecconi M, De Backer D, Antonelli M, Beale R, Bakker J, Hofer C, Jaeschke R, Mebazaa A, Pinsky MR, Teboul JL, Vincent JL, Rhodes A. Consensus on circulatory shock and hemodynamic monitoring. Task force of the European Society of Intensive Care Medicine. Intensive Care Med. 2014 Dec;40(12):1795-815. doi: 10.1007/s00134-014-3525-z. Epub 2014 Nov 13. PMID 25392034
- [Background] Biais M, Larghi M, Henriot J, de Courson H, Sesay M, Nouette-Gaulain K. End-Expiratory Occlusion Test Predicts Fluid Responsiveness in Patients With Protective Ventilation in the Operating Room. Anesth Analg. 2017 Dec;125(6):1889-1895. doi: 10.1213/ANE.0000000000002322. PMID 28742783
- [Derived] Messina A, Lionetti G, Foti L, Bellotti E, Marcomini N, Cammarota G, Bennett V, Saderi L, Sotgiu G, Della Corte F, Protti A, Monge Garcia MI, Romagnoli S, Cecconi M. Mini fluid chAllenge aNd End-expiratory occlusion test to assess flUid responsiVEness in the opeRating room (MANEUVER study): A multicentre cohort study. Eur J Anaesthesiol. 2021 Apr 1;38(4):422-431. doi: 10.1097/EJA.0000000000001406. PMID 33399372